CLINICAL TRIAL: NCT04701047
Title: Prospective Observational Study with Patient Reported Outcome Measures (PROM) for the Treatment of Vaginal Prolapse: Pessary Vs. Surgery
Brief Title: Prospective Observational Prolapse Study
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08720-ADP
Record Dates: First submitted 2020-12-02; First posted 2021-01-08 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse | interventions — Pessaries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- pessary: Vaginal prolapse being treated by pessary
  Interventions: Device: vaginal pessary
- surgery: Vaginal prolapse being treated by surgical repair
  Interventions: Procedure: Vaginal prolapse surgery

INTERVENTIONS:
Device: vaginal pessary — insertion and follow up of a vaginal pessary
  Groups: pessary
Procedure: Vaginal prolapse surgery — surgery and follow up after vaginal prolapse surgery
  Groups: surgery

SUMMARY:
The rationale of the study is to investigate the results of a prolapse treatment in adult women with a vaginal prolapse. The investigators will investigate this by taking questionnaires in women undergoing a surgical prolapse repair and in women that are being treated by a vaginal pessary. The objective is to compare the results of the different methods with each other and to observe the evolution of the symptoms in patients undergoing surgery or pessary use. The investigators would also like to discover existing problems in pessary use and adverse effects.

DETAILED DESCRIPTION:
The rationale of the study is to investigate the results of a prolapse treatment in adult women with a vaginal prolapse. The investigators will investigate this by taking questionnaires in women undergoing a surgical prolapse repair and in women that are being treated by a vaginal pessary. The objective is to compare the results of the different methods with each other and to observe the evolution of the symptoms in patients undergoing surgery or pessary use. The investigators would also like to discover existing problems in pessary use and adverse effects.

The questionnaires that will be used are the PFDI-20 (pelvic floor distress inventory), PFIQ-7 (pelvic floor impact questionnaire), PISQ-9 (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire) and a custom-made questionnaire to further investigate the behavior towards pessary use of our patients and the adverse effects they are dealing with. The questionnaires will be taken before the treatment has started, 6 weeks post treatment start, one-year post treatment start, two years post treatment start and 5 years post treatment start. A POP-Q (Pelvic Organ Prolapse Quantification) investigation will be performed to estimate the degree of vaginal prolapse before the start of the treatment. Since clinical follow up is not necessarily needed after one year for the women who undergo surgery, their questionnaires will be taken via telephone or e-mail. For women that are being treated with pessaries the investigators will also take our custom-made questionnaire at 4 and 8 months after starting the treatment.

The investigators would like to recruit 100 women for this study, older than 18 years old who have not undergone a previous treatment with a pessary or surgery for vaginal prolapse. Another exclusion criterium are women who still have a child wish and women who have contraindications for surgery. The investigators will also exclude women who don't speak Dutch or women who cannot give a written consent.

The investigators hypothesize that woman being treated with one year of pessary use are overall not having more symptoms than woman that underwent a surgery. The investigators hypothesize that woman being treated with five years of pessary use are overall having less symptoms than woman that underwent a surgery.

ELIGIBILITY:
Inclusion Criteria:

* women with a symptomatic vaginal prolapse
* older than 18 years

Exclusion Criteria:

* under 18 years old
* undergone a previous treatment with a pessary or surgery for vaginal prolapse
* contra-indications for surgery or pessary use
* active or passive child wish
* not able to understand the Dutch language
* not able to give a written consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research population will include women above the age of 18 years old who consult the department of urology or the department of gynaecology at the university hospital of Ghent with symptoms of vaginal prolapse. The patients will be recruited by their attending physician. There will be no exclusion on the degree of vaginal prolapse. All symptomatic prolapses will be included in this study. Exclusion criteria will be having undergone a previous treatment with a pessary or surgery for vaginal prolapse, contraindications for surgery or pessary use, active of passive child wish, not able to understand the Dutch language and not able to give a written consent.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pelvic Floor Disability Index (PFDI-20) | Baseline, 6 weeks, one year, two years, five years
  Change in scores on the short-form version of the Pelvic Floor Distress Inventory (PFDI). It is a health-related quality of life questionnaire for women with pelvic floor conditions to fill out.
Change in pelvic floor impact questionnaire (PFIQ-7) | Baseline, 6 weeks, one year, two years, five years
  Change in scores on the shortened version of the Pelvic Floor Impact Questionnaire (PFIQ). It is a health-related quality of life questionnaire for women with pelvic floor conditions to fill out.
Change in Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | Baseline, 6 weeks, one year, two years, five years
  Change in scores on the short form of the PISQ-31 that evaluates sexual function in women with urinary incontinence and/or pelvic organ prolapse

SECONDARY OUTCOMES:
Subjective self-reported satisfaction scores for pessary use as measured via a custom-made Likert scale questionnaire | 4 months after start of therapy
  Study participants are asked how satisfied they are with their pessary use at 4 months after the initiation of pessary use. Participants can choose one of five graded answers on the Likert scale:
  5 Very satisfied 4 satisfied 3 neutral 2 unsatisfied
  1 very unsatisfied
Subjective self-reported satisfaction scores for pessary use as measured via a custom-made Likert scale questionnaire | 8 months after start of therapy
  Study participants are asked how satisfied they are with their pessary use at 8 months after the initiation of pessary use. Participants can choose one of five graded answers on the Likert scale:
  5 Very satisfied 4 satisfied 3 neutral 2 unsatisfied
  1 very unsatisfied
Self-reported behavior and patient preferences towards pessary use via a custom-made questionnaire | 4 months after initiation of therapy
  frequency of pessary use, subjective reasons why not to wear a pessary and alternative treatment considerations as assessed by open-ended and yes or no type questions
Self-reported behavior and patient preferences towards pessary use via a custom-made questionnaire | 8 months after initiation of therapy
  frequency of pessary use, subjective reasons why not to wear a pessary and alternative treatment considerations as assessed by open-ended and yes or no type questions
Subjective self-reported adverse effects of pessary use as measured via a custom-made questionnaire | 4 months after initiation of therapy
  Participants will be asked if they experienced side effects that they feel has been caused by pessary use via a custom-made questionnaire: The most commonly anticipated answers have been listed with the option of patients describing other potential adverse events (shown below):
  * No side effects
  * It feels uncomfortable
  * It gives an itchy/burning sensation
  * More vaginal discharge
  * Other……….
Subjective self-reported adverse effects of pessary use as measured via a custom-made questionnaire | 8 months after initiation of therapy
  Participants will be asked if they experienced side effects that they feel has been caused by pessary use via a custom-made questionnaire: The most commonly anticipated answers have been listed with the option of patients describing other potential adverse events (shown below):
  * No side effects
  * It feels uncomfortable
  * It gives an itchy/burning sensation
  * More vaginal discharge
  * Other……….

OTHER OUTCOMES:
Amount of pessaries tried before current pessary | 4 months after initiation of therapy
  Number of pessaries that are being fitted before finding a suitable one via a custom made questionnaire.
Amount of pessaries tried before current pessary | 8 months after initiation of therapy
  Number of pessaries that are being fitted before finding a suitable one via a custom made questionnaire.
Duration of the pessary consultation | 4 months after initiation of therapy
  Duration of a pessary consultation in minutes.
Duration of the pessary consultation | 8 months after initiation of therapy
  Duration of a pessary consultation in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Tjalina Hamerlynck, Principal Investigator — UZ Gent; Steven Weyers, Principal Investigator — UZ Gent; Van Wessel Steffi, Study Director — UZ Gent; Abosi Appeadu Kessewa, Study Chair — UZ Gent; Decalf Veerle, Study Chair — UZ Gent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided